CLINICAL TRIAL: NCT03267121
Title: A Non-randomized Phase II Study of Apatinib and Tegafur Gimeracil Oteracil Induction Chemotherapy in Locally Advanced Squamous Cell Carcinoma of Head and Neck
Brief Title: A Study of Apatinib and Tegafur Gimeracil Oteracil in Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Guopei Zhu, M.D., Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017HNRT002
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2022-07

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: head and neck cancer; Apatinib; Tegafur Gimeracil Oteracil; induction chemotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — apatinib; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental): Apatinib Mesylate Tablets and Tegafur Gimeracil Oteracil Potassium Capsules administered as a daily oral treatment
  Interventions: Drug: Apatinib Mesylate Tablets; Drug: Tegafur Gimeracil Oteracil Potassium Capsules

INTERVENTIONS:
Drug: Apatinib Mesylate Tablets — 500 mg qd.p.o. every day for 21 days as a cycle
  Other Names: Aitan
Drug: Tegafur Gimeracil Oteracil Potassium Capsules — 25mg/㎡ bid p.o. every day for 14 days as a cycle
  Other Names: Aiyi; S-1

SUMMARY:
This is a non-randomized, phase II, open label study of apatinib mesylate tablets plus tegafur gimeracil oteracil potassium capsules induction chemotherapy in locally advanced squamous cell carcinoma of head and neck patients who were judged surgically unresectable or appropriate for non-surgical definitive therapy.The primary purpose of this study is to evaluate the efficacy of apatinib mesylate tablets plus tegafur gimeracil oteracil potassium capsules in locally advanced squamous cell carcinoma of head and neck

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed SCCHN or poorly differentiated or undifferentiated cancer of the head and neck.
2. Measurable disease.
3. All primary sites are eligible excluding nasopharyngeal.
4. Surgically unresectable and/or refuse surgery; Note: surgical unresectability will be defined as the combination of the treating surgeon's judgment of unresectability plus one of the following objective criteria:

   Encasement of tumor or nodes to the carotid artery or ¾ encasement of the carotid artery.

   Involvement of prevertebral musculature Invasion of the bone of the skull base Need for glossectomy or extensive glossal resection where functional outcome is considered unacceptable to surgeon or patient Involvement of the cervical spine Severe, unacceptable functional deficit that would result from any proposed definitive surgical resection.
5. ECOG performance status 0-1
6. Age > or = 18 years. Men and women are eligible for participation.
7. Must have acceptable organ and marrow function as defined below. Laboratory tests should be completed within 14 days prior to registration:

   Absolute Neutrophil Count (ANC) > or = 1,500/mm3 Platelets > or = 100,000/mm3 Hemoglobin (Hgb) > 9g/dL Total bilirubin < or = 1.5mg/dL Albumin > 2.5 g/dL Aspartate aminotransferase (AST)/Alanine Aminotransferase (ALT) < or = 2.5 times institutional upper limit of normal, alkaline phosphatase < 2.5 x upper limit of normal, glomerular filtration rate (GFR) > 30 mL/min (by standard Cockcroft and Gault formula or measured via 24 hour urine collection)
8. Patients must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients with poor-controlled arterial hypertension (systolic pressure ≥ 140 mmHg and/or diastolic pressure ≥ 90 mm Hg) despite standard medical management;
2. Suffered from grade II or above myocardial ischemia or myocardial infarction, uncontrolled arrhythmias (including QT interval male ≥ 450 ms, female ≥ 470 ms). Grade III-IV cardiac insufficiency according to New York Heart Association (NYHA) criteria or echocardiography check: left ventricular ejection fraction (LVEF)<50%;
3. Patients who have had prior allergic reaction to Apatinib and Tegafur Gimeracil Oteracil;
4. The subject has had another active malignancy within the past five years except for cervical cancer in site, in situ carcinoma of the bladder or non-melanoma carcinoma of the skin;
5. Clinically significant and uncontrolled major medical conditions including but not limited to: active uncontrolled infection, symptomatic congestive heart failure, Unstable angina pectoris or cardiac arrhythmia, psychiatric illness/ social situation that would limit compliance with study requirements; any medical condition, which in the opinion of the study investigator places the subject at an unacceptably high risk for toxicities;
6. Patients undergoing therapy with other investigational agents.
7. Women who are pregnant or breastfeeding;
8. Patients with any other concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (CR+PR) | 9 weeks
  Objective Response Rate as defined by RECIST 1.1 after induction chemotherapy followed by definitive chemoradiation. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response (OR) = CR + PR.

SECONDARY OUTCOMES:
Number of Participants With at Least One Grade 3-4 Toxicity | 9 weeks
  Toxicity will be assessed according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.
Progression Free Survival | 3 years
  Rate of Progression Free Survival (Time to death or progression defined by imaging of target lesions via CT or MRI scan post induction chemotherapy and chemoradiotherapy)
Overall Survival | 3 years
  Rate of Progression Free Survival (Time to death post induction chemotherapy and chemoradiotherapy)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai ninth people's hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jiang W, Li R, Zhang L, Dou S, Ye L, Shao Z, Wu S, Dong M, Li J, Zhu G. Efficacy and feasibility of Apatinib and S-1 as a novel oral induction therapy in locally advanced head and neck squamous cell carcinoma: an exploratory phase 2 open-label, single-arm trial. Front Oncol. 2023 May 12;13:1072538. doi: 10.3389/fonc.2023.1072538. eCollection 2023. PMID 37251944
- See also: Related Info — https://www.frontiersin.org/journals/oncology/articles/10.3389/fonc.2023.1072538/full